CLINICAL TRIAL: NCT01187303
Title: Ofatumumab in Relapsed Nodular Lymphocyte Predominant Hodgkin Lymphoma (NLPHL)
Brief Title: Ofatumumab in Nodular Lymphocyte Predominant Hodgkin Lymphoma (NLPHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1432
Record Dates: First submitted 2010-08-19; First posted 2010-08-24 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Relapsed NLPHL
MeSH Terms: conditions — Hodgkin Disease | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ofatumumab — 300 mg/m2 d1 week 1 1000mg/m2 d1 week 2-8

SUMMARY:
The purpose of this trial is to determine the efficacy of ofatumumab in patients with relapsed nodular lymphocyte predominant Hodgkin lymphoma (NLPHL).

ELIGIBILITY:
Inclusion Criteria:

* relapsed nodular lymphocyte predominant hodgkin lymphoma
* age 18 - 75
* review of diagnosis by experienced pathologist
* no major organ dysfunction

Exclusion Criteria:

* classical hodgkin lymphoma
* CD20 antibody treatment within the last 6 months prior enrollment
* chronic or current infectious disease requirering systemic antibiotics
* other past or current malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 12 months after end of treatment

SECONDARY OUTCOMES:
duration of response | 12 months after end of treatment
Progression free survival | 12 months after end of treatment
adverse events | 12 months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, MD, Principal Investigator — University of Cologne
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- See also: Homepage of the German Hodgkin Study Group — http://ww.ghsg.org